CLINICAL TRIAL: NCT06145490
Title: Adenosine Receptors from Genes to Behavior: Neurobehavioral Correlates of Caffeine on Anxiety, Avoidance, Decision-Making and Interoception in Healthy Individuals and Panic Disorder.
Brief Title: Neurobehavioral Correlates of Caffeine on Anxiety, Avoidance and Interoception in Healthy Individuals and Panic Disorder.
Acronym: BINCAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2023-02915-02
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Panic Disorder; Healthy
MeSH Terms: conditions — Panic Disorder | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: The study entails two sessions with a cross-over design. Participants will be randomized to start with either the caffeine condition or the placebo condition.
  The study includes two arms: (a) participants with Panic Disorder (anticipated n = 50) and (b) Healthy controls (anticipated n = 50). Both arms (Panic Disorder and Healthy controls) will complete both conditions with the two sessions (caffeine and placebo condition) in randomized order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Panic Disorder (Other): Participants will be randomized to start with either the caffeine condition or the placebo condition. Participants will complete session 2 with the other condition (condition not allocated to in session 1).
  Interventions: Dietary Supplement: Caffeine; Drug: Placebo
- Healthy controls (Other): Participants will be randomized to start with either the caffeine condition or the placebo condition. Participants will complete session 2 with the other condition (condition not allocated to in session 1).
  Interventions: Dietary Supplement: Caffeine; Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine — Caffeine capsule 250 mg, oral intake
Drug: Placebo — Placebo capsule, oral intake

SUMMARY:
The current study is a placebo-controlled, double-blind, randomized controlled study using a cross-over design, including Healthy Controls (HC) and participants with Panic Disorder (PD).

The primary aim of the study is to investigate the neural correlates and behavioral effects of caffeine (versus placebo), and its impact on emotional reactivity, decision-making, and interoception, and compare the effects in individuals with PD vs HCs. Subjective anxiety and the occurrence of panic attacks will also be measured. Multimodal neuroimaging methods, such as structural and functional MRI, will be used to address the aims of the study.

Emotional reactivity, emotional decision-making and interoception will be measured with experimental tasks in a 7 Tesla (7T) magnetic resonance (MR) scanner, jointly with measures of skin conductance, heart rate, respiratory rate, and self-reported ratings of anxiety and interoception.

Emotional reactivity will be assessed using emotional and neutral faces. Emotional decision-making will be assessed with an approach-avoidance conflict task. Changes in interoception (bodily sensation, such as pulse and respiration) will be explored using a task in which participants are asked to focus on their breathing or an external stimulus. Caffeine effects on brain resting-state activity will also be assessed. All tasks will be conducted while in the 7T MR scanner.

A secondary aim of the study is to examine the impact of genetic variability in the adenosine A2A receptor (ADORA2A) genotype (e.g., rs5751876 T/T) on the effects of caffeine (vs placebo), as ADORA2A genotype has previously been associated with elevated caffeine-induced anxiety.

DETAILED DESCRIPTION:
Given the novelty of the intended study and the lack of previous neuroimaging and emotion-related behavioral studies on caffeine effects in HCs and PD, analyses will be exploratory without directed hypotheses.

It is intended to conduct between-group analyses (HCs vs PD) in the two conditions (caffeine versus placebo), as well as within-group analyses in HCs and PD separately. Between-group analyses will also be conducted between individuals with different ADORA2A genotypes.

ELIGIBILITY:
Inclusion Criteria:

* Panic Disorder group (PD): Primary diagnosis of Panic Disorder.
* Healthy control group (HCs): No current or history of psychiatric disorders.
* All participants (PD and HCs): Weekly caffeine consumption ≤ 300 mg.

Exclusion Criteria:

* Weekly caffeine consumption ≥ 300 mg.
* Thoracic or head surgery, or any other surgery or metallic implanted devices not compatible with the safety standards for 7T MR scanner.
* History of severe psychiatric disorder (e.g., schizophrenia).
* Somatic or neurological conditions (e.g., hypertension and heart condition).
* Ongoing treatment with psychotropic medication or treatment with psychotropic medication which has been discontinued within 2 months.
* Other ongoing treatments that may confound the results.
* Current drug or alcohol abuse/dependency.
* Habitual nicotine use.
* Uncorrected visual or hearing impairment.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Task-related BOLD fMRI signal | Session 1 (day 1)
  Task-related BOLD (blood-oxygen-level-dependent) fMRI (functional magnetic resonance imaging) signal will be collected through a 7T MR scanner, starting approximately 30 minutes after oral intake of caffeine or placebo pill. Tasks: Emotional reactivity, Approach-Avoidance Conflict Task, Interoception, Resting-state fMRI.
Task-related BOLD fMRI signal | Session 2 (day 2; minimum of 36 hours after session/day 1)
  Task-related BOLD (blood-oxygen-level-dependent) fMRI (functional magnetic resonance imaging) signal will be collected through a 7T MR scanner, starting approximately 30 minutes after oral intake of caffeine or placebo pill. Tasks: Emotional reactivity, Approach-Avoidance Conflict Task, Interoception, Resting-state fMRI.
Self-reported anxiety | Session 1 (day 1)
  Anxiety will be assessed before capsule intake (either caffeine or placebo), 20 minutes after intake, after each task, and during the interoception task measured with self-reported ratings, on a scale from 0-100 (0= no anxiety - 100= extreme anxiety).
Self-reported anxiety | Session 2 (day 2; minimum of 36 hours after session/day 1)
  Anxiety will be assessed before capsule intake (either caffeine or placebo), 20 minutes after intake, after each task, and during the interoception task measured with self-reported ratings, on a scale from 0-100 (0= no anxiety - 100= extreme anxiety).
Self-reported interoceptive awareness | Session 1 (day 1)
  Interoceptive awareness will be assessed before capsule intake (either caffeine or placebo), 20 minutes after intake, after each task in the MR scanner, and during the interoception task, measured with self-reported ratings on a scale from 0-100 (0= no awareness - 100= extreme awareness).
Self-reported interoceptive awareness | Session 2 (day 2; minimum of 36 hours after session/day 1)
  Interoceptive awareness will be assessed before capsule intake (either caffeine or placebo), 20 minutes after intake, after each task in the MR scanner, and during the interoception task, measured with self-reported ratings on a scale from 0-100 (0= no awareness - 100= extreme awareness).
Self-reported interoceptive functional impairment | Session 1 (day 1)
  Interoceptive functional impairment will be assessed before capsule intake (either caffeine or placebo), 20 minutes after intake, after each task, and during the interoception task, measured with self-reported ratings on a scale from 0-100 (0= no impairment - 100= extreme impairment).
Self-reported interoceptive functional impairment | Session 2 (day 2; minimum of 36 hours after session/day 1)
  Interoceptive functional impairment will be assessed before capsule intake (either caffeine or placebo), 20 minutes after intake, after each task, and during the interoception task, measured with self-reported ratings on a scale from 0-100 (0= no impairment - 100= extreme impairment).
Skin conductance responses (SCR) | Session 1 (day 1)
  Skin conductance responses will be used to assess emotional reactivity at the physiological level to emotional stimuli vs neutral stimuli (faces).
Skin conductance responses (SCR) | Session 2 (day 2; minimum of 36 hours after session/day 1)
  Skin conductance responses will be used to assess emotional reactivity at the physiological level to emotional stimuli vs neutral stimuli (faces).
Occurrence of panic attacks | Session 1 (day 1)
  The occurrence of panic attacks will be assessed according to the Diagnostic Statistical Manual (DSM-5) criteria for panic attacks and will be coded dichotomous as "present" or "not present".
Occurrence of panic attacks | Session 2 (day 2; minimum of 36 hours after session/day 1)
  The occurrence of panic attacks will be assessed according to the Diagnostic Statistical Manual (DSM-5) criteria for panic attacks and will be coded dichotomous as "present" or "not present".

SECONDARY OUTCOMES:
Structural brain data, T1-w sMRI | Session 1 (day 1)
  Structural brain changes will be analyzed through T1-weighted sMRI (structural magnetic resonance imaging).
Structural brain data, T1-w sMRI | Session 2 (day 2; minimum of 36 hours after session/day 1)
  Structural brain changes will be analyzed through T1-weighted sMRI (structural magnetic resonance imaging).
Heart rate variability | Session 1 (day 1)
  Heart rate variability (HRV) will be assessed by using a 7T MR-compatible heart rate band, during the whole MR scanner time.
Heart rate variability | Session 2 (day 2; minimum of 36 hours after session/day 1)
  Heart rate variability (HRV) will be assessed by using a 7T MR-compatible heart rate band, during the whole MR scanner time.
Respiratory rate | Session 1 (day 1)
  Respiratory or breathing rates will be assessed during the whole MR scanner time.
Respiratory rate | Session 2 (day 2; minimum of 36 hours after session/day 1)
  Respiratory or breathing rates will be assessed during the whole MR scanner time.

OTHER OUTCOMES:
Expectancy ratings | Session 1 (day 1)
  Participants will be asked to report if they believed they received placebo or caffeine and how certain they are on a scale from 0-100% before capsule intake and after completing the MR-session.
Expectancy ratings | Session 2 (day 2; minimum of 36 hours after session/day 1)
  Participants will be asked to report if they believed they received placebo or caffeine and how certain they are on a scale from 0-100% before capsule intake and after completing the MR-session.
Panic Disorder Severity Scale (PDSS) | 1-7 days prior to session 1 (internet)
  PDSS is a self-reported questionnaire that assesses the severity of Panic Disorder; range 0-28, higher scores indicating more severe symptoms.
Body Sensations Questionnaire (BSQ) | 1-7 days prior to session 1 (internet)
  BSQ assesses body sensations present during aversive situations; range 17-85, higher scores indicating higher levels of body sensations.
Multidimensional Assessment of Interoceptive Awareness (MAIA-2) | 1-7 days prior to session 1 (internet)
  MAIA-2 is an 8-scale state-trait questionnaire with 37 items to measure multiple dimensions of interoception by self- report. The score of each scale is the the average of the items on each scale. Higher mean scores indicate higher levels of the measured dimensions (Noticing, Not-Distracting, Not-Worrying, Attention Regulation, Emotional Awareness,Self-Regulation, Body Listening, and Trust) on a scale from 0-5 (0=never- 5=always), respectively.
Anxiety Sensitivity Index (ASI) | 1-7 days prior to session 1 (internet)
  ASI assesses anxiety sensitivity; range 0-64, higher scores indicating higher anxiety sensitivity.
Spielberger State-Trait Anxiety Inventory (STAI-T) | 1-7 days prior to session 1 (internet)
  STAI-T is a self-rated questionnaire assessing trait anxiety; range 20-80, higher scores represent higher levels of trait anxiety.
Caffeine Expectancy Questionnaire (CaffEQ) | 1-7 days prior to session 1 (internet)
  CaffEQ is a self-rated questionnaire that assesses expected effect of caffeine intake.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Frick, PhD, Principal Investigator — Uppsala University, Department of Medical Sciences, Psychiatry
Locations (2):
- Sweden (2):
  - National 7T Facility - Lunds universitet, Lund
  - Uppsala University, Department of Medical Sciences, Psychiatry, Uppsala

IPD SHARING:
Plan to Share IPD: No